CLINICAL TRIAL: NCT04686331
Title: Diagnostic and Prognostic Accuracy of Surfactant Protein D, Krebs Von Den Lungen, and Chitinase-3-like Protein 1 (YKL-40 ) in the Initial Investigation of Patients With Suspected Pneumonia
Brief Title: Accuracy of Lung Injury Biomarkers in the Initial Investigation of Patients With Suspected Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-12d-2020
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Community-acquired Pneumonia
Keywords: surfactant protein D; Krebs von den Lungen; YKL-40 C; pneumonia; lung injury; diagnostic markers; prognostic markers; emergency department
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Lung Injury; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected CAP: All patients admitted to the emergency department with suspected community-acquired pneumonia (CAP) assessed by the receiving physician
  Interventions: Diagnostic Test: Biomarkers for pneumonia

INTERVENTIONS:
Diagnostic Test: Biomarkers for pneumonia — Blood samples will be collected by a medical laboratory technologist and transferred to the local laboratory for analysis of surfactant protein D, Krebs von den Lungen (KL-6), and YKL-40. Laboratory staff will be blinded to participant diagnosis and outcome. None of the biomarkers will be available to the treating physician.
  * Diagnostic test of surfactant protein D - will be quantified using enzyme-linked immunosorbent assay (ELISA)-based analysis
  * Diagnostic test of KL-6: will be quantified using enzyme-linked immunosorbent assay (ELISA)-based analysis
  * Diagnostic test of YKL-40 - will be quantified using enzyme-linked immunosorbent assay (ELISA)-based analysis

SUMMARY:
The aim of this study is to investigate the diagnostic and prognostic value of surfactant protein D, Krebs von den Lungen (KL-6), and Chitinase-3-like protein 1 (YKL-40) in the initial investigation of patients hospitalized with suspected pneumonia. This to improve the diagnosis of pneumonia, contribute to a more rapid and accurate antibiotic treatment, and assess disease severity to predict short-term and long-term mortality in community-acquired pneumonia patients.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is one of the most common infection diseases in the emergency department (ED). Diagnosis of pneumonia is challenging as symptoms are often weak and nonspecific and the current methods for focal and etiological diagnosis have low sensitivity and specificity and often deliver results after the antibiotic treatment decision has been made.

The abundant and restricted expression of surfactant protein D (SP-D) within the lung makes this protein a specific marker for lung disease. Krebs von den Lungen-6 (KL-6) is expressed in the lung and is a diagnostic and prognostic marker of interstitial lung disease. The inflammatory glycoprotein Chitinase-3-like protein 1 commonly known as YKL-40 is associated with severity of interstitial lung disease. The value of these lung injury markers for diagnosing pneumonia needs further investigation.

The investigators hypothesize that surfactant protein D, Krebs von den Lungen (KL-6), and Chitinase-3-like protein 1 (YKL-40) have an impact on diagnosing, prognosis, and treatment of patients with verified CAP.

The objectives of the study are:

* To investigate the diagnostic accuracy of surfactant protein D, Krebs von den Lungen (KL-6), and Chitinase-3-like protein 1 (YKL-40) in the diagnosis of CAP
* To identify the prognostic value surfactant protein D, Krebs von den Lungen (KL-6), and Chitinase-3-like protein 1 (YKL-40) in relation to adverse events in patients with verified CAP

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of APN assessed by the receiving physician at the ED

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients with suspected Acute pyelonephritis (APN) from three emergency departments (EDs) in the Region of Southern Denmark (Hospital Sønderjylland, Hospital Lillebælt, Odense University Hospital)
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Verified and non-verified community acquired pneumonia (CAP) | 2 months after patient discharge
  The decision of whether patients admitted with suspicion of CAP actually has a final diagnosis of CAP is based on a combination of all findings during admission. The verification of diagnosis requires human handling, interpretation and judgment. Therefore, in this study, an expert panel will define the reference standard for the diagnosis CAP. The expert panel consists of two independent consultants from the emergency department with significant experience in emergency medicine and acute infections. They will individually determine whether or not the patient admitted suspected with CAP actually had this diagnosis. The final diagnosis will be based on all available relevant information from the patient medical record including HR-CT of lungs. A standardized template will be used. Disagreement will be discussed until a consensus is reached.

SECONDARY OUTCOMES:
Intensive care unit treatment | within 60 days from admission to the emergency department
  transfer to ICU during current admission (binary outcome)
Length of stay | within 60 days from current admission to the emergency department
  days spent in hospital during current admission
the number of participants who died within 30 days | within 30 days from arrival day
  binary - 30-days mortality
The number of participants who died within 90 days | within 90 days from arrival day
  binary - 90-days mortality
Readmission | within 30 days from day of discharge
  binary
In-hospital mortality | within 60 days from admission to the emergency department
  binary

OTHER OUTCOMES:
Bacteriuria | urine collected within 4 hours of arrival to emergency department
  Binary outcome defined by microbiologist on urine culture analysis
Diagnostic capabilities of Ultra low-dose computer thermography for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for ultra low-dose computer thermography for pneumonia.
Diagnostic capabilities of lung ultrasound for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for lunge ultrasound for pneumonia.
Diagnostic capabilities of chest x-ray for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for chest x-ray for pneumonia
Level of infection markers | blood collected with 4 hours of arrival to emergency department
  Concentration of serum procalcitonin, CRP and suPAR
CURB-65 severity score | within 4 hours from admission
  Confusion of new onset, Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL), respiratory rate of 30 breaths per minute or greater, blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less and age 65 or older. The score stratify patients to groups 1 (mild pneumonia), 2 (moderate pneumonia) and 3-5 (severe pneumonia).
Pneumonia severity index (PSI) | within 4 hours from admission
  Risk classes to predict the severity of pneumonia. Scores are given based on demographics, comorbidity, clinical measurements and physical Exam Findings (<70 = Risk Class II, 71-90 = Risk Class III, 91-130 = Risk Class IV, >130 = Risk Class V)
Microbial agents | results within 7 days from sputum sample collection
  Microbial agents (bacteria and viruses) identified in standard culture, PCR and multiplex PCR. Sputum or tracheal secretion samples are collected within 1 hour from patient admission.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishikawa N, Hattori N, Yokoyama A, Kohno N. Utility of KL-6/MUC1 in the clinical management of interstitial lung diseases. Respir Investig. 2012 Mar;50(1):3-13. doi: 10.1016/j.resinv.2012.02.001. Epub 2012 Mar 8. PMID 22554854
- [Background] Sorensen GL. Surfactant Protein D in Respiratory and Non-Respiratory Diseases. Front Med (Lausanne). 2018 Feb 8;5:18. doi: 10.3389/fmed.2018.00018. eCollection 2018. PMID 29473039
- [Background] Furuhashi K, Suda T, Nakamura Y, Inui N, Hashimoto D, Miwa S, Hayakawa H, Kusagaya H, Nakano Y, Nakamura H, Chida K. Increased expression of YKL-40, a chitinase-like protein, in serum and lung of patients with idiopathic pulmonary fibrosis. Respir Med. 2010 Aug;104(8):1204-10. doi: 10.1016/j.rmed.2010.02.026. Epub 2010 Mar 27. PMID 20347285